CLINICAL TRIAL: NCT06492148
Title: Effect of Myofascial Release Technique on Central Sensitization, Myofascial Trigger Point and Menstrual Symptoms in Women With Primary Dysmenorrhea: Sham-Controlled, Randomized Double-Blind Study
Brief Title: Myofascial Release Technique in Women With Primary Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, BEYZA YAZGAN DAĞLI, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023 - 1577
Record Dates: First submitted 2024-06-11; First posted 2024-07-09 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Dysmenorrhea Primary; Central Sensitisation; Myofascial Trigger Point Pain; Menstrual Discomfort; Myofascial Release
Keywords: myofascial release; trigger point; Central sensitization; Dysmenorrhea; sham
MeSH Terms: conditions — Myofascial Pain Syndromes; Dysmenorrhea | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release Group (Active Comparator): The technique known as myofascial release, also referred to as cross-hand release, will be applied to 7 regions. Among these regions are the lateral abdominal wall (right and left), the lower abdomen with the opposite side medial thigh (right and left crossed), the thoracolumbar fascia (bilateral), and the lumbosacral region. In the cross-hand technique, hands will be gently placed on the specified regions and directions. The release of the barriers of the tissue under the hands will be ensured, and the technique will be applied until a wave or oscillation is felt. A myofascial release technique with an optimal duration of 5 minutes will be applied to each region. The total treatment time will be 35 minutes.
  Interventions: Other: Myofascial Release
- Sham- Myofascial Release Group (Sham Comparator): The hands of the researcher applying the technique will be positioned on the same regions as the myofascial release technique, with only the palms lightly touching for the same duration. However, there will be no intervention aimed at applying pressure or opening tissue barriers. The total sham treatment time will be 35 minutes.
  Interventions: Other: Sham-Myofascial Release

INTERVENTIONS:
Other: Myofascial Release — The myofascial release technique is a widely used manual therapy method characterized by low-load, prolonged mechanical forces applied to manipulate the myofascial complex, aiming to restore optimal length, alleviate pain, and improve function.
  Arms: Myofascial Release Group
Other: Sham-Myofascial Release — The hands of the researcher applying the technique will be placed in the same areas as the myofascial release technique, with only the palms in light contact for the same duration. However, no intervention will be made to create any pressure or open the tissue barrier.
  Arms: Sham- Myofascial Release Group

SUMMARY:
It has been found that women with dysmenorrhea have active trigger points, particularly in the rectus abdominis, oblique abdominal muscles, quadratus lumborum, and paraspinal muscles. The myofascial release technique is a widely used manual therapy method characterized by the application of low-load, long-duration mechanical forces to manipulate the myofascial complex. This technique aims to restore optimal length, alleviate pain, and improve function. This study aims to examine the effect of the myofascial release technique on central sensitization, myofascial trigger points, and menstrual symptoms in women with primary dysmenorrhea.

DETAILED DESCRIPTION:
During the evaluation period, the participants' musculoskeletal pain threshold and tolerance will be measured using an algometer, about trigger points on the identified muscles (rectus abdominis, quadratus lumborum, erector spinae, and tibialis anterior). A total of 40 women, aged 18-40, diagnosed with primary dysmenorrhea by a gynecologist, will be included in the study. The initial assessment of the participants will be conducted on their most painful days. Participants will be randomized into two groups: the myofascial release technique group (study group) and the placebo myofascial release technique group (control group). The interventions will be conducted over 10 sessions during one menstrual cycle, and all evaluations will be repeated after the treatment period. The study will be conducted as a double-blind trial, ensuring that both the evaluators and the patients are blind to the group assignments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Primary Dysmenorrhea according to the Primary Dysmenorrhea Consensus Guide,
* Having regular menstruation in the last 6 months (28±7 days)
* Those who had menstrual pain between 40 mm and 100 mm according to the Visual Analogue Scale (VAS) in the last 6 months

Exclusion Criteria:

* Diagnosed with Secondary Dysmenorrhea,
* Having given birth,
* Those with serious gastrointestinal, urogynecological, or autoimmune diseases or other chronic pain syndromes,
* Undergoing urogynecological surgery,
* Those who are pregnant or suspected of pregnancy,
* Those who use analgesics or non-pharmacological agents other than NSAIDs for menstrual pain,
* Those using intrauterine or oral contraceptives,
* Those taking extra supplements such as magnesium, which may affect treatment

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Pain Pressure Threshold | Baseline (First menstruation cycle)
  Trigger points in specific muscles (rectus abdominis, paraspinal muscles, quadratus lumborum, gluteus maximus) will be determined. Then, it will be applied to the trigger points with the Baseline brand algometer in accordance with standard procedures and the pressure will be increased by 30 kPa/s.
Pain Pressure Threshold | through study completion, an average of 3 months
  Trigger points in specific muscles (rectus abdominis, paraspinal muscles, quadratus lumborum, gluteus maximus) will be determined. Then, it will be applied to the trigger points with the Baseline brand algometer in accordance with standard procedures and the pressure will be increased by 30 kPa/s.
Central Sensitization | Baseline (First menstruation cycle)
  Pain threshold will be measured with an algometer at a certain point of the tibialis muscle.
Central Sensitization | through study completion, an average of 3 months
  Pain threshold will be measured with an algometer at a certain point of the tibialis muscle.
Menstrual pain intensity | Baseline (First menstruation cycle)
  Menstrual pain intensity will be determined by a 10 cm Visual Analog Scale ranging from zero (no pain at all) to 10 (worst pain I have ever felt). Higher scores mean worse conditions. Participants will be asked to mark the severity of pain they felt in the first 3 days of their last menstrual bleeding on 3 separate lines.
Menstrual pain intensity | through study completion, an average of 3 months
  Menstrual pain intensity will be determined by a 10 cm Visual Analog Scale ranging from zero (no pain at all) to 10 (worst pain I have ever felt). Higher scores mean worse conditions. Participants will be asked to mark the severity of pain they felt in the first 3 days of their last menstrual bleeding on 3 separate lines.

SECONDARY OUTCOMES:
Menstrual Attitude | Baseline (First menstruation cycle)
  Menstrual Attitude Scale will be used to evaluate symptoms related to menstruation. High scores indicate a high awareness of menstruation.
Menstrual Attitude | through study completion, an average of 3 months
  Menstrual Attitude Scale will be used to evaluate symptoms related to menstruation. High scores indicate a high awareness of menstruation.
Health-related quality of life | Baseline (First menstruation cycle)
  Short Form (SF-36) will be used to evaluate individuals' general health-related quality of life. SF-36 is a 36-question survey that evaluates functionality and well-being and consists of 8 subscales. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Higher scores indicate a better quality of life.
Health-related quality of life | through study completion, an average of 3 months
  SF-36 will be used to evaluate individuals' general health-related quality of life. SF-36 is a 36-question survey that evaluates functionality and well-being and consists of 8 subscales. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Higher scores indicate a better quality of life.
Anxiety | Baseline (First menstruation cycle)
  State and Trait Anxiety Scale is a self-assessment inventory that evaluates anxiety and consists of 40 items.
Anxiety | through study completion, an average of 3 months
  State and Trait Anxiety Scale is a self-assessment inventory that evaluates anxiety and consists of 40 items.
The Body Awareness | Baseline (First menstruation cycle)
  The Body Awareness Questionnaire will be used to evaluate changes in individuals' body awareness. The questionnaire consists of 18 items and 4 subscales (predicting body reactions, sleep-wake cycle, predicting the onset of the disease, paying attention to changes in body processes).
The Body Awareness | through study completion, an average of 3 months
  The Body Awareness Questionnaire will be used to evaluate changes in individuals' body awareness. The questionnaire consists of 18 items and 4 subscales (predicting body reactions, sleep-wake cycle, predicting the onset of the disease, paying attention to changes in body processes).

CONTACTS AND LOCATIONS:
Overall Officials: Beyza Yazgan Dagli, Principal Investigator — Gazi University
Locations (1):
- Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No